CLINICAL TRIAL: NCT04127305
Title: Drug Monitoring of Antiinfectives in Critically Ill Patients Receiving Extracorporeal Life Support - a Prospective Observational Pilot Study
Brief Title: Drug Monitoring in Critically Ill Patients During Extracorporeal Life Support
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Elisabeth H. Adam, Principal investigator, Goethe University
Other Study IDs: Drug Monitoring during ECMO
Record Dates: First submitted 2019-10-12; First posted 2019-10-15 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Drug Monitoring of Antiinfectives in Critically Ill Patients Receiving Extracorporeal Life Support
Keywords: drug monitoring; antiinfectives; intensive care; ECMO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- VA ECMO: Patients will be included at the beginning of VA ECMO therapy within 24-48h after start of an antiinfective therapy
  Interventions: Other: No Intervention
- VA EMCO + RRT: Patients with RRT will be included at the beginning of VA ECMO therapy within 24-48h after start of an antiinfective therapy
  Interventions: Other: No Intervention
- VV ECMO: Patients will be included at the beginning of VV ECMO therapy within 24-48h after start of an antiinfective therapy
  Interventions: Other: No Intervention
- VV ECMO + RRT: Patients with RRT will be included at the beginning of VV ECMO therapy within 24-48h after start of an antiinfective therapy
  Interventions: Other: No Intervention
- Control: Patients will be included within 24-48h after start of an antiinfective therapy
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
About 70% of critically ill patients require antiinfective therapy. Optimal antibiotic dosing is key to improve patient survival, reduce toxic effects and minimise the emergence of bacterial resistance. There is a growing body of evidence demonstrating the existence of significant changes in pharmacokinetics (PK) in intensive care patients, particularly those with extracorporeal therapy (extracorporeal membrane oxygenation (ECMO), continuous renal replacement therapy (CRRT)). To characterize the effects of extracorporal therapy for critically ill patients, we designed a prospective pilot observational study using a drug monitoring to derive relevant effects of extracorporeal therapy and clinical patient characteristics for the treatment with meropenem, teicoplanin, linezolid, piperacillin/tazobactam, levofloxacin and acyclovir.

DETAILED DESCRIPTION:
About 70% of critically ill patients require antiinfective therapy. Optimal antibiotic dosing is key to improve patient survival, reduce toxic effects and minimise the emergence of bacterial resistance. However, there is a growing body of evidence demonstrating the existence of significant changes in pharmacokinetics (PK) in intensive care patients, particularly those with extracorporeal therapy (extracorporeal membrane oxygenation (ECMO), continuous renal replacement therapy (CRRT)). Existing antiinfectivedosing regimens assume a "normal" PK; currently there are no evidence-based antiinfective dosing guidelines for critically ill patients available. The current recommendations of the Paul-Ehrlich Society and the Surviving Sepsis Campaign therefore recommend explicitly appliance of a therapeutic drug monitoring (TDM) for intensive care patients to individually adjust dosing and to avoid potential over- or underdosing. To characterize the effects of extracorporal therapy for critically ill patients, we designed a prospective pilot observational study using a drug monitoring. Six antiinfectives (meropenem, teicoplanin, linezolid, piperacillin / tazobactam, levofloxacin and aciclovir) will be investigated as index substances for the various antiinfective groups. A total of 100 patients, divided into 5 groups of 20 patients, will be examined in this study: 1. venovenous (vv)-ECMO, 2. venoarterial (va)-ECMO, 3. vv-ECMO + CRRT, 4. va-ECMO + CRRT, 5. control group. Sampling for determination of trough and peak levels of the study substances will take place during the different dosing intervals. Patients will be included at the beginning of ECMO therapy within 24-48h after start of an antiinfective therapy with at least one of the index-substances; observation period will be a total of 5 days. The collected data will be analyzed to identify covariates associated with changes in PK for the 6 different antiinfectives in critically ill patients receiving extracorporeal therapy. Using the comprehensive data set collected, the pharmacokinetic profile of the 6 antiinfectives as well as other influencing factors will be constructed to assess the need for dose adjustment of antiinfective agents in these patients. This prospective observational trial addresses the current knowledge deficiency with the aim to derive relevant effects of extracorporeal therapy and clinical patient characteristics for the treatment with meropenem, teicoplanin, linezolid, piperacillin/tazobactam, levofloxacin and acyclovir. With these relevant results, adapted dosing of antiinfectives can probably be improved in critically ill patients with extracorporeal therapy in future.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Informed consent
* Clinical infection indicated for intravenous therapy with at least one of the following index anti-infectives: meropenem, teicoplanin, linezolid, piperacillin/tazobactam, levofloxacin and/oraciclovir
* Application of an ECLS procedure with an expected duration of at least five days

Exclusion Criteria:

* Pregnancy
* Massive Hemorrhage

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: critically ill patients with extracorporeal heart or lung support and possibly CRRT
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of antiinfective agents | 12 months
  pharmacokinetic profile of 6 antiinfectives (meropenem, teicoplanin, linezolid, piperacillin / tazobactam, levofloxacin and aciclovir) as well as other influencing factors will be constructed to assess the need for dose adjustment of antiinfective agents

CONTACTS AND LOCATIONS:
Locations (1):
- Universital Hospital Frankfurt / Main, Frankfurt am Main, Deutschland, Germany

IPD SHARING:
Plan to Share IPD: No